CLINICAL TRIAL: NCT03812666
Title: Inflammatory Biomarkers In Stroke - Discovery Phase
Brief Title: Search for Biomarkers of Infection and Inflammation in Patients With Acute Stroke.
Acronym: IBIS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jakob Ström (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Sponsor-Investigator, Jakob Ström, Jakob Ström, MD, PhD, resident of neurology and Associate Professor, Region Örebro County
Organization: Region Örebro County (Other)
Other Study IDs: 247991; 2018/288 (Other: Regional ethical review board Uppsala)
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute; Pneumonia, Bacterial
Keywords: Stroke; Pneumonia; Biomarkers; Infection
MeSH Terms: conditions — Stroke; Pneumonia, Bacterial; Pneumonia; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Daily blood samples for 7 days as well as a 90-day follow-up blood sample will be stored in a biobank for later analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe stroke: Patients with severe (defined as NIHSS score of > 10) acute stroke, either ischemic or hemorrhagic. (n= 150)
- Moderately stroke: Patients with moderately severe (defined as NIHSS score of > 5 but < 11) acute stroke, either ischemic or hemorrhagic. (n= 25)
- Mild stroke: Patients with mild (defined as NIHSS score of <6) acute stroke, either ischemic or hemorrhagic. (n= 25)

SUMMARY:
This study will look for new biomarkers of infection and evaluate current biomarkers of infection in stroke patients. Patients with acute stroke will be monitored with daily blood samples for seven days and by clinical examination to detect infections for 10 days.

DETAILED DESCRIPTION:
Rationale: Stroke is one of the leading causes of death globally, and infections after stroke contribute to a large part of the stroke-related mortality. The current study, which has a prospective, observational design, constitutes the second phase out of four in the Inflammatory Biomarkers In Stroke (IBIS) project, of which the overall goal is to enable early treatment of post-stroke infections.

Aim: To develop a combined clinical and molecular biological signature for early detection of pneumonia in patients with stroke.

Design: Prospective nested case control study

Methods:Patients (n=200) with acute stroke will be monitored with clinical examinations for ten days and by daily blood samples for seven days. When cases of pneumonia have been established, samples and examination results from days preceding overt pneumonia will be compared to samples from similar patients that did not develop pneumonia.

Outcome: Using proteomic and metabolomic methods, novel markers of upcoming pneumonia after stroke will be sought. Such laboratory markers will be combined with current biomarkers (such as C-reactive protein and procalcitonin) and data from clinical examinations, with the aim of constructing a biological signature that enables early detection of pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and radiology consistent with acute cerebral infarction or atraumatic intracerebral hemorrhage.
* National Institutes of Health Stroke Scale (NIHSS) ≤5; mild stroke (n=25), NIHSS ≤10 and ≥ 6; moderate stroke (n=25) or NIHSS ≥ 11; severe stroke (n=150)
* Onset of symptoms less than 48 hours before first study blood sampling.

Exclusion Criteria:

* Symptoms and radiology consistent with acute cerebral infarction but full reversal of symptoms within 24 hours of onset. (i.e. transient ischemic attack, TIA)
* Hemoglobin less than 90 g/l.
* Ongoing inflammatory disease, such as rheumatoid arthritis or active inflammatory bowel disease.
* Inability to undergo MRI scan (only patients with NIHSS ≤10 will be excluded by this criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients admitted to Örebro University hospital will be consecutively offered enrollement. The sample is weighted to include more patients with severe stroke (defined as NIHSS ≥ 11) than with moderate (NIHSS ≤10 and ≥ 6) or mild (NIHSS ≤5) stroke. The purpose of this is to ensure that a high proportion of participants will contract pneumonia since patients with a more severe stroke have a higher risk of pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Novel biomarkers of pneumonia | The day before pneumonia onset.
  The study will analyze a broad expanse of potential biomarkers, including known markers of infection such as c-reactive protein, procalcitonin and increased respiratory frequency as well as novel markers that will be pursued using proteomic and metabolomic methods. Those that are significantly associated with upcoming pneumonia will be selected. Biomarkers will be evaluated by the area under the curve for the receiver operating characteristic (AUC-ROC).
A combined clinical and molecular biological signature for early detection of pneumonia | The day before pneumonia onset.
  By combining novel (found using proteomic and metabolomic methods) and current biomarkers (such as c-reactive protein, procalcitonin and increased respiratory frequency) with data from clinical examinations, a biological signature that enables early detection of pneumonia will be constructed.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Ström, MD, PhD, Principal Investigator — Region Örebro County
Locations (1):
- Örebro University Hospital, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sjolin K, Royter B, Forgo B, Aulin J, Kultima K, Lindback J, Strom JO, Burman J. Plasma Profiles of Neuroglial Injury Biomarkers after Ischemic Stroke. Transl Stroke Res. 2025 Dec;16(6):2185-2194. doi: 10.1007/s12975-025-01380-y. Epub 2025 Sep 3. PMID 40900222